CLINICAL TRIAL: NCT00811044
Title: Regulation of Hepatic Insulin Extraction:Alterations of Insulin Secretion in Subjects With Genetic Variants That Determine Risk for Non-Insulin Dependant Diabetes Mellitus
Brief Title: Regulation of Hepatic Insulin Extraction
Acronym: RHIE
Status: Withdrawn | Type: Observational
Why Stopped: PI, Dr. K. Polonsky has moved to the University of Chicago.
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Chicago (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00-0589; 5R01DK031842-26 (NIH)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Diabetes
Keywords: diabetes; genetics; oral glucose tolerance testing; family history of diabetes; gestational diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples are collected for Glucose & various human peptide measurements and DNA. As peptide assay evolves, specimens may be re-tested.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Entry: This group is just entering the study and will need to be genotyped.
- Affected: This group has been genotyped and has the gene undergoing study at that time.
- Control: This group has been genotyped and does not have the gene currently under study.

SUMMARY:
* This study is in the area of Type 2 diabetes and genetics
* Healthy Volunteers and those with mild type 2 diabetes may be eligible to participate
* This study is searching for genes that may affect the body's processing/digestion of glucose/sugar

DETAILED DESCRIPTION:
This study is looking at the genetic influences of type 2 diabetes. It also is investigating the various gastric hormones including but not limited to: insulin, C-peptide, GIP, GLP, & Xenin.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* non-diabetic
* diabetes controlled with diet or with pills
* no family history of diabetes
* family history of type 2 diabetes
* personal history of gestational diabetes

Exclusion Criteria:

* < 18 or > 65 years of age
* medications that affect glucose (sugar) levels
* kidney disease
* liver disease
* heart/cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers & otherwise healthy diabetic volunteers (do not require insulin for glucose control).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2000-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Genes affecting the development of Type 2 diabetes will be identified | 1 year

SECONDARY OUTCOMES:
Any differences between genetic groups in the metabolism of glucose/sugar will be studied to the extent that the data allow | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Polonsky, MD, Principal Investigator — Washington University School of Medicine